CLINICAL TRIAL: NCT02516813
Title: An Open Label, Phase Ia/Ib Trial of the DNA-PK Inhibitor MSC2490484A in Combination With Radiotherapy in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Trial of MSC2490484A, an Inhibitor of a DNA-dependent Protein Kinase, in Combination With Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100036-002; 2015-000673-12 (EudraCT Number)
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors
Keywords: M3814; Advanced solid tumors; DNA-PK Inhibitor; Radiotherapy; Chemotherapy
MeSH Terms: interventions — peposertib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Phase 1a (Arm A): M3814 Capsule (100 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative radiotherapy (RT) received 100 milligrams (mg) of M3814 as capsule orally once daily on fraction day (FD) 6 in combination with RT (3 Gray [Gy] x 10, 5 fractions per week [F/W]).
  Interventions: Drug: M3814 100 mg; Radiation: Fractionated RT
- Phase 1a (Arm A): M3814 Capsule (200 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative RT received 200 mg of M3814 as capsule orally once daily on FD 6 in combination with RT (3 [Gy] x 10, 5 F/W).
  Interventions: Drug: M3814 200 mg; Radiation: Fractionated RT
- Phase 1a (Arm A): M3814 Capsule (300 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative RT received 300 mg of M3814 as capsule orally once daily on FD 6 in combination with RT (3 [Gy] x 10, 5 F/W).
  Interventions: Drug: M3814 300 mg; Radiation: Fractionated RT
- Phase 1a (Arm A): M3814 Capsule (400 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative RT received 400 mg of M3814 as capsule orally once daily on FD 6 in combination with RT (3 [Gy] x 10, 5 F/W).
  Interventions: Drug: M3814 400 mg; Radiation: Fractionated RT
- Phase 1a (Arm A): M3814 Tablet (100 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative RT received 100 mg of M3814 as tablet orally once daily for 2 consecutive weeks in combination with RT (3 Gy x 10, 5 F/W).
  Interventions: Drug: M3814 100 mg; Radiation: Fractionated RT
- Phase 1a (Arm A): M3814 Tablet (200 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative RT received 200 mg of M3814 as tablet orally once daily for 2 consecutive weeks in combination with RT (3 Gy x 10, 5 F/W).
  Interventions: Drug: M3814 200 mg; Radiation: Fractionated RT
- Phase 1a (Arm A): M3814 Tablet (300 mg) + RT (Experimental): Participants with locally advanced disease (any tumor or metastases including lymphomas) localized in the head and neck region or thorax that was not amenable to surgical therapy, or with standard systemic therapy with an indication for palliative RT received 300 mg of M3814 as tablet orally once daily for 2 consecutive weeks in combination with RT (3 Gy x 10, 5 F/W).
  Interventions: Drug: M3814 300 mg; Radiation: Fractionated RT
- Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT (Experimental): Participants with local/locally advanced squamous cell carcinoma of the head and neck (SCCHN) received 50 mg of M3814 as capsule orally once daily on FD 6 in combination with fractionated RT (2 Gy x 33 to 35 fractions; 5 F/W) and Cisplatin twice at a dose of 100 milligrams per square meter (mg/m^2) or weekly at a dose of 40 (mg/m^2).
  Interventions: Drug: M3814 50 mg; Radiation: Fractionated RT; Drug: Cisplatin
- Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) received 100 mg of M3814 as tablet orally once daily for 7 consecutive weeks in combination with fractionated RT (2 Gy X 33 to 35 fractions; 5 F/W) and Cisplatin twice at a dose of 100 mg/m^2 or weekly at a dose of 40 (mg/m^2).
  Interventions: Radiation: Fractionated RT; Drug: Cisplatin
- Ancillary cPoP: M3814 Capsule (100 mg) + RT (Experimental): Participants with at least 2 (sub)cutaneous tumor/metastases of any type (at least 2 centimeters [cm] apart) with an indication for single high dose-palliative RT were included and received single oral dose of M3814 capsule at a dose of 100 mg on Day 2, prior 1.5 hours start of RT and a single high dose of RT (10-25 Gy) on Lesion 1 on Day 1 and on Lesion 2 on Day 2.
  Interventions: Drug: M3814 100 mg; Radiation: Fractionated RT
- Ancillary cPOP: M3814 Capsule (200 mg) + RT (Experimental): Participants with at least 2 (sub)cutaneous tumor/metastases of any type (at least 2 cm apart) with an indication for single high dose-palliative RT were included and received single oral dose of M3814 capsule at a dose of 200 mg on Day 2, prior 1.5 hours start of RT and a single high dose of RT (10-25 Gy) on Lesion 1 on Day 1 and on Lesion 2 on Day 2.
  Interventions: Drug: M3814 200 mg; Radiation: Fractionated RT
- Ancillary cPOP: M3814 Capsule (400 mg) + RT (Experimental): Participants with at least 2 (sub)cutaneous tumor/metastases of any type (at least 2 cm apart) with an indication for single high dose-palliative RT were included and received single oral dose of M3814 capsule at a dose of 400 mg on Day 2, prior 1.5 hours start of RT and a single high dose of RT (10-25 Gy) on Lesion 1 on Day 1 and on Lesion 2 on Day 2
  Interventions: Drug: M3814 400 mg; Radiation: Fractionated RT

INTERVENTIONS:
Drug: M3814 100 mg — Participants received 100 mg of M3814 as capsule or tablet orally once daily.
  Other Names: Peposertib; MSC2490484A
  Arms: Ancillary cPoP: M3814 Capsule (100 mg) + RT; Phase 1a (Arm A): M3814 Capsule (100 mg) + RT; Phase 1a (Arm A): M3814 Tablet (100 mg) + RT
Drug: M3814 200 mg — Participants received 200 mg of M3814 as capsule or tablet orally once daily.
  Other Names: Peposertib; MSC2490484
  Arms: Ancillary cPOP: M3814 Capsule (200 mg) + RT; Phase 1a (Arm A): M3814 Capsule (200 mg) + RT; Phase 1a (Arm A): M3814 Tablet (200 mg) + RT
Drug: M3814 300 mg — Participants received 300 mg of M3814 as capsule or tablet orally once daily.
  Other Names: Peposertib; MSC2490484
  Arms: Phase 1a (Arm A): M3814 Capsule (300 mg) + RT; Phase 1a (Arm A): M3814 Tablet (300 mg) + RT
Drug: M3814 400 mg — Participants received 400 mg of M3814 as capsule or tablet orally once daily.
  Other Names: Peposertib; MSC2490484
  Arms: Ancillary cPOP: M3814 Capsule (400 mg) + RT; Phase 1a (Arm A): M3814 Capsule (400 mg) + RT
Drug: M3814 50 mg — Participants received 100 mg of M3814 as capsule orally once daily.
  Other Names: Peposertib; MSC2490484
  Arms: Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT
Radiation: Fractionated RT — Participants received fractionated palliative RT (3 Gray [Gy] * 10 in Arm A and 2 Gy * 33 to 35, 5 fractions per week [F/W]) in Arm B and received a single high dose of RT (10-25 Gy) capsule on Day 1 given on Lesion 1 and a single high dose of RT (10-25 Gy) on Day 2 given on Lesion 2 in ancillary CPoP part.
Drug: Cisplatin — Participants received Cisplatin twice at a dose of 100 mg/m^2 or weekly at a dose of 40 mg/m^2.
  Arms: Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT; Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT

SUMMARY:
M3814 was an investigational drug that is being evaluated for the treatment of participants with locally advanced tumors. The main purposes of this study was to determine the safety, the tolerability and the efficacy of M3814 in combination with radiotherapy and in combination with chemoradiotherapy (Radiotherapy + cisplatin).

ELIGIBILITY:
Inclusion Criteria:

* Phase Ia part: advanced solid tumors or metastases including lymphoma localized in the head and neck region or thorax with an indication for fractionated palliative RT (Arm A); or treatment-naïve SCCHN eligible for fractionated curatively intended RT with concurrent cisplatin (Arm B)
* Phase Ib part: treatment-naïve Stage III A/B NSCLC not eligible for surgical resection or concurrent chemoradiation (Arm A expansion cohort) or treatment-naïve SCCHN eligible for fractionated curatively intended RT with concurrent cisplatin (Arm B expansion cohort)
* Ancillary cPoP Part: any tumor with at least 2 (sub)cutaneous tumor/metastases at least 2 cm apart which are RT naïve with an indication for high dose palliative RT
* Availability of archival tumor material, either as a block or slides (Phase Ia and Ib). If no archival material is available then a fresh biopsy should be taken
* Willing to have tumor biopsies collected in Ancillary cPoP
* Measurable or evaluable disease by RECIST v1.1 (not required for ancillary cPoP part of the study)
* Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 1
* Life expectancy of ≥ 3 months (Phase Ia, Arm A) or ≥ 6 months (Phase Ia, Arm B and Phase Ib)
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy.

Exclusion Criteria:

* Chemotherapy, immunotherapy, hormonal therapy, biologic therapy, or any other anticancer therapy or investigational medicinal product (IMP) within 28 days of first trial drug intake for Phase Ia subjects, and any prior therapy for Phase Ib subjects. For subjects with rapidly growing tumors localized in the head and neck region or thorax where the treating physician cannot wait for 28 days, inclusion may take place if there is no residual toxicity from previous treatment (maximum CTCAE Grade 1)
* Prior RT to the same region within 12 months (Phase Ia, Arm A; subjects with tumors localized in the head and neck region or thorax) or at any time previously (Phase Ia, Arm B; treatment-naïve subjects with SCCHN and Phase Ib; treatment-naïve subjects with Stage III A/B NSCLC or SCCHN)
* Extensive prior RT on ≥30% of bone marrow reserve as judged by the investigator or prior bone marrow/stem cell transplantation within 5 years before trial start.
* Poor vital organ functions defined as:

  * Bone marrow impairment as evidenced by hemoglobin <10.0 g/dL, neutrophil count <1.0 × 109/L, platelets <100 × 109/L
  * Renal impairment as evidenced by serum creatinine >1.5 × upper limit of normal (ULN)
  * Liver function abnormality as defined by total bilirubin >1.5 × ULN or aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >2.5 × ULN (except for subjects with liver involvement, who can have AST/ALT >5 × ULN)
* History of difficulty swallowing, malabsorption or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the IMP, use of percutaneous endoscopic gastrostomy (PEG) tubes
* Significant cardiac conduction abnormalities, including a history of long QTc syndrome and/or pacemaker, or impaired cardiovascular function such as New York Heart Association classification score >2.
* Subjects currently receiving (or unable to stop using prior to receiving the first dose of trial drug) medications or herbal supplements known to be potent inhibitors of cytochrome P450 (CYP)3A or CYP2C19 (must stop at least 1 week prior), potent inducers of CYP3A or CYP2C19 (must stop at least 3 weeks prior), or drugs mainly metabolized by CYP3A with a narrow therapeutic index (must stop at least one day prior).
* Subjects currently receiving H2-blocker or proton pump inhibitors (or unable to stop at least 5 days prior to the first treatment).
* If the planned radiation field includes any part of the esophagus and the subject has symptoms of ongoing esophagitis, the subject is not eligible, unless an esophageal endoscopy rules out the presence of esophagitis
* Subjects where more than 10% of the total esophagus volume receives more than 50% of the prescribed RT dose

Main exclusion criteria for Ancillary Clinical Proof-of-Principle Part:

* History of difficulty swallowing, malabsorption or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the IMP
* History of any other significant medical disease such as major gastric or small bowel surgery, recent drainage of significant volumes of ascites or pleural effusion (as per Investigator's judgement) or a psychiatric condition that might impair the subject's well-being or preclude full participation in the trial
* Subjects currently receiving (or unable to stop using prior to receiving the first dose of study drug) medications or herbal supplements known to be potent inhibitors of CYP3A or CYP2C19 must stop at least 1 week prior to taking MSC2490484A. Subjects receiving potent inducers of CYP3A or CYP2C19 must stop at least 3 weeks prior to taking MSC2490484A. Those receiving drugs mainly metabolized by CYP3A with a narrow therapeutic index as judged by the Investigator (and after optional consultation with the Sponsor) must stop at least one day prior to taking MSC2490484A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (26):
- United States (9):
  - Research site, Fresno, California
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Research site, Billings, Montana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Research site, Houston, Texas
  - Research site, Tacoma, Washington
- Research site, Leuven, Belgium
- Denmark (2):
  - Rigshospitalet - PARENT, Copenhagen
  - Herlev Hospital - PARENT, Herlev
- Germany (9):
  - Research site, Freiburg im Breisgau, Baden-Wurttemberg
  - Charite Research Organisation GmbH - Phase - I Unit of Hematology and Oncology, Berlin
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Essen - Westdeutsches Tumorzentrum, Essen
  - Universitaetsklinikum Heidelberg - RadioOnkologie und Strahlentherapie, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel - Klinik für diagnostische Radiologie, Kiel
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz - Klinik und Poliklinik fuer Radiologie, Mainz
  - Klinikum Mannheim GmbH Universitaetsklinikum - Parent, Mannheim
  - Universitaetsklinikum Tuebingen - Medizinische Klinik I, Tübingen
- Netherlands (2):
  - Research site, Amsterdam
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
- Research site, Oslo, Norway
- Karolinska universitetssjukhuset - Solna - Radiumhemmet (onkologi), Solna, Sweden
- Universitaetsspital Zuerich - Parent, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=100036-002
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Participant First Visit (FPFV): 15 September 2015; Last Participant last Visit (LPLV): 19 November 2021
Pre-assignment Details: The study was planned to be conducted in 3 parts: Phase Ia (dose escalation), Phase Ib (dose expansion) and Ancillary clinical proof-of-principle (cPoP). Phase Ib part of the study was never initiated due to early discontinuation as per sponsor's decision.
Period: Overall Study
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Started | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3 | 3 | 3 | 1
Completed | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT | Total
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3 | 3 | 3 | 1 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 2 | 3 | 2 | 4 | 7 | 2 | 2 | 1 | 0 | 31
  >=65 years | 3 | 1 | 1 | 4 | 3 | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2 | 2 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 13
  Male | 6 | 2 | 3 | 4 | 4 | 2 | 4 | 8 | 2 | 1 | 2 | 1 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 8
  Not Hispanic or Latino | 7 | 2 | 2 | 5 | 5 | 3 | 4 | 4 | 3 | 3 | 3 | 1 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  White | 7 | 3 | 3 | 5 | 6 | 3 | 5 | 5 | 3 | 2 | 3 | 1 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a (Arm A): Number of Participants Who Experienced at Least One Dose-limiting Toxicity (DLT) According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: DLT: any Grade (Gr) greater than or equal to (>=) 3 nonhematologic adverse event (AE)/any Gr>=4 hematologic AE that is related to any of study treatments and occurs during the DLT period of 5 weeks (Phase Ia, Arm A) after the first dose of M3814. Following are considered as DLTs: Gr3 thrombocytopenia with medically concerning bleeding; Febrile neutropenia; Any toxicity/study treatment-related adverse event (TEAE) that, in opinion of Safety Monitoring Committee (SMC), is of potential clinical significance such that further dose escalation would expose participants to unacceptable risk; Any toxicity related to study treatments that causes participant to receive less than 80 percent (%) of the planned RT dose; Evidence of study treatment-related hepatocellular injury for > 3 days.
Time Frame: Time from first dose of study treatment up to 5 weeks
Population: Dose-Escalation Analysis Set included all participants treated in dose-escalation cohorts who received at least 80% of the M3813 and RT planned dose and completed the DLT period (5 weeks after the start of RT) or who experienced a DLT during DLT period regardless of the amount of treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT
Number analyzed (Participants) | 7 | 3 | 2 | 6 | 6 | 3 | 6
Participants | 1 | 0 | 2 | 3 | 1 | 0 | 3

2. Primary Outcome: Phase 1a (Arm B): Number of Participants Who Experienced at Least One Dose-limiting Toxicity (DLT) According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: DLT: any Grade (Gr) greater than or equal to (>=) 3 nonhematologic AE/any Gr>=4 hematologic AE that is related to any of study treatments and occurs during the DLT period of 12 weeks (Phase Ia, Arm B) after the first dose of M3814. Following are considered as DLTs: Gr3 thrombocytopenia with medically concerning bleeding; Febrile neutropenia; Any toxicity/study treatment-related adverse event (TEAE) that, in opinion of Safety Monitoring Committee (SMC), is of potential clinical significance such that further dose escalation would expose participants to unacceptable risk; Any toxicity related to study treatments that causes participant to receive less than 80 percent (%) of the planned RT dose; Any toxicity related to study treatments leading to an interruption of RT longer than 1 week in Arm B; Evidence of study treatment-related hepatocellular injury for > 3 days.
Time Frame: Time from first dose of study treatment up to 12 weeks
Population: Dose-Escalation Analysis Set included all participants treated in dose-escalation cohorts who received at least 80% of the M3814 and RT planned dose and completed the DLT period (12 weeks after the start of RT) or who experienced a DLT during DLT period regardless of the amount of treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3
Participants | 2 | 2

3. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Grade Greater Than or Equal to (>=) 3 Treatment-Emergent Adverse Events (TEAEs) According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily have a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious AEs and non-serious AEs. As per NCI-CTCAE v4.03, Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death. Number of participants with Grade >=3 TEAEs were reported.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: Safety analysis set included all participants who received at >= 1 administration of study intervention (either M3814 or RT).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3
Participants | 2 | 3 | 3 | 3 | 3 | 0 | 5 | 8 | 3

4. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Shifts From Baseline to Worst Post-Baseline Grade in Hematology Parameters According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTC v4.03)
Description: Number of participants with shifts from Baseline values (Grade 0/1/2) to worst post-baseline values (Grade 1/2/3/4) were reported as per NCI-CTCAE, v4.03 graded from Grade 1 to 5. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death. Shifts in hematology parameter (hemoglobin low, leukocytes low, lymphocytes low, neutrophil count decreased, and platelet count decreased) were reported.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3
Participants
  Hemoglobin low: Grade 0 to Grade 1 | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 3 | 0
  Hemoglobin low: Grade 0 to Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Hemoglobin low: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin low: Grade 1 to Grade 2 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0
  Hemoglobin low: Grade 1 to Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes low: Grade 0 to Grade 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1
  Leukocytes low: Grade 0 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
  Leukocytes low: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Leukocytes low: Grade 1 to Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes low: Grade 0 to Grade 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Lymphocytes low: Grade 0 to Grade 2 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 0
  Lymphocytes low: Grade 0 to Grade 3 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 4 | 1
  Lymphocytes low: Grade 0 to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Lymphocytes low: Grade 1 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocytes low: Grade 1 to Grade 3 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Lymphocytes low: Grade 1 to Grade 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Lymphocytes low: Grade 2 to Grade 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocytes low: Grade 2 to Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased: Grade 0 to Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  Neutrophil count decreased: Grade 0 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Neutrophil count decreased: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophil count decreased: Grade 1 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets count decreased: Grade 0 to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets count decreased: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Shifts From Baseline to Worst Post-Baseline Grade in Biochemistry Parameters According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Number of participants with shifts from Baseline values (Grade 0/1/2) to worst post-baseline values (Grade 1/2/3/4) were reported as per NCI-CTCAE, v4.03 graded from Grade 1 to 5. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death. Shifts in biochemistry parameter (phosphate low, potassium low, sodium low, alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, blood bilirubin increased, glucose high, glucose low, albumin low and creatinine increased) were reported.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: Safety analysis set included all participants who received at >= 1 administration of study intervention (either M3814 or RT). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 2 | 6 | 6 | 3 | 6 | 8 | 3
Participants
  Phosphate low: Grade 0 to Grade 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
  Phosphate low: Grade 0 to Grade 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1
  Phosphate low: Grade 1 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Phosphate low: Grade 2 to Grade 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Potassium low: Grade 0 to Grade 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1
  Potassium low: Grade 0 to Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Sodium low: Grade 0 to Grade 1 | 2 | 2 | 1 | 0 | 2 | 0 | 3 | 4 | 1
  Alanine aminotransferase: Grade 0 to Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
  Alkaline phosphatase: Grade 0 to Grade 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 0
  Aspartate aminotransferase: Grade 0 to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
  Blood bilirubin increased: Grade 0 to Grade 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Glucose high: Grade 0 to Grade 1 | 3 | 0 | 0 | 3 | 2 | 2 | 1 | 0 | 0
  Glucose high: Grade 0 to Grade 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose high: Grade 1 to Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Glucose high: Grade 1 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Glucose high: Grade 2 to Grade 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
  Glucose low: Grade 0 to Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Albumin low: Grade 0 to Grade 1 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 0
  Albumin low: Grade 0 to Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Albumin low: Grade 1 to Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Creatinine increased: Grade 0 to Grade 1 | 5 | 3 | 1 | 5 | 5 | 3 | 5 | 6 | 1
  Creatinine increased: Grade 0 to Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine increased: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine increased: Grade 1 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Markedly Abnormal Vital Sign Measurements
Description: Vital sign assessments included assessments of heart rate, blood pressure, body weight and body temperature. Abnormal vital sign measurement was decided by Investigator. Number of participants with markedly abnormal vital sign measurements were reported.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Shifts From Normal Baseline to Abnormal Post-baseline in Electrocardiogram (ECG)
Description: Electrocardiograms (ECG) was obtained after the participant has been in a supine position for at least 5 minutes. ECG parameters included heart rate, atrial ventricular conduction, QR and QT intervals (including QTcF), and possible arrhythmias. Any ECG finding that was judged by the investigator as a abnormal (worsening) compared with a baseline value was considered an adverse event. Number of participants with shifts from normal baseline values to abnormal post-baseline values in ECG were reported.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0

8. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Confirmed Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: Confirmed BOR was defined as best response of any of complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from date of randomization until disease progression. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD: defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. CR or PR must be confirmed by a subsequent tumor assessment, at least 4 weeks after initial documentation of CR or PR.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: Full analysis set included all participants who received at >= 1 administration of study intervention (either M3814 or RT).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
  Partial response (PR) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Stable disease (SD) | 5 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 0
  Progressive disease (PD) | 1 | 0 | 1 | 1 | 5 | 2 | 3 | 0 | 0
  Not Evaluable | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0

9. Secondary Outcome: Phase 1a (Arm A and Arm B): Number of Participants With Unconfirmed Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: Unconfirmed BOR was defined as unconfirmed best response of any of complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from date of randomization until disease progression. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD: defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 6 | 8 | 3
Participants
  Complete response (CR) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 0
  Partial response (PR) | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3
  Stable disease (SD) | 3 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 0
  Progressive disease (PD) | 1 | 0 | 1 | 1 | 5 | 2 | 3 | 0 | 0
  Not Evaluable | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0

10. Secondary Outcome: Phase 1a (Arm A and Arm B): Median Percent Change From Baseline in Tumor Size Measurement According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: The tumor size was defined as the sum of the longest diameters for the target lesions. The sum of lesion diameters was calculated using RECIST v1.1 and was assessed by Investigator.
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Population: as for outcome 8
Measure: Median (Full Range); unit: percentage change
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 2 | 2 | 5 | 6 | 3 | 5 | 6 | 3
percentage change | -25.81 [-88.06 to 0.00] | -41.29 [-60.00 to -22.58] | -3.95 [-7.89 to 0.00] | -21.95 [-82.14 to 10.61] | -20.84 [-81.25 to -2.13] | -9.52 [-28.0 to 9.82] | -40.00 [-100 to 6.98] | -100 [-100 to -61.11] | -52.78 [-71.43 to -43.55]

11. Secondary Outcome: Phase 1a (Arm A and Arm B): Maximum Plasma Concentration (Cmax) of M3814 After Single Dose
Description: Cmax was taken directly from the observed concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: Pharmacokinetic analysis set: all participants who received at least the first dose of the treatment (either M3814 or RT) and provided >= 3 valid post-dose concentration points within 6 hours (0-6 hours inclusive). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and number analyzed= participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 5 | 8 | 3
nanogram per milliliter (ng/mL)
  Fraction Day 1 | 378 (91.2) | 1260 (12.5) | 515 (94.5) | 1630 (62.9) | 724 (77.8) | 799 (37.9) | 2260 (112.6) | 173 (87.2) | 599 (34.2)
  Fraction Day 6: number analyzed (Participants) | 6 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 314 (150.4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 840 (20.8) |  |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

12. Secondary Outcome: Phase 1a (Arm A and Arm B): Time to Reach Maximum Plasma Concentration (Tmax) of M3814 After Single Dose
Description: tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: Pharmacokinetic analysis set included all participants who received at least the first dose of the treatment (either M3814 or RT) and provided >= 3 valid post-dose concentration points within 6 hours (0-6 hours inclusive). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed"= participants evaluable at specified timepoints.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 5 | 8 | 3
hours
  Fraction Day 1 | 2.03 [1.00 to 4.03] | 2.05 [1.00 to 2.18] | 3.98 [1.00 to 4.00] | 2.03 [0.95 to 3.75] | 1.18 [0.42 to 4.00] | 1.17 [1.00 to 2.15] | 1.00 [0.83 to 4.48] | 2.34 [0.98 to 4.08] | 1.00 [0.98 to 2.05]
  Fraction Day 6: number analyzed (Participants) | 6 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 0.93 [0.50 to 4.02] | NA [NA to NA] — Median and full range was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 2.01 [2.00 to 2.15] |  |  | NA [NA to NA] — Median and full range was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

13. Secondary Outcome: Phase 1a (Arm A and Arm B): Area Under the Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of M3814 After Single Dose
Description: AUC0-24 of M3814 was defined as the area under the concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 3 | 5 | 7 | 3
hour*nanogram per milliliter (h*ng/mL)
  Fraction Day 1: number analyzed (Participants) | 4 | 3 | 3 | 3 | 6 | 3 | 5 | 7 | 3
  Fraction Day 1 | 2310 (52.2) | 7580 (49.5) | 4950 (71.1) | 14700 (56.1) | 2490 (191.6) | 3800 (71.7) | 14100 (97.7) | 969 (52.1) | 2890 (119.8)
  Fraction Day 6: number analyzed (Participants) | 5 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 915 (133.0) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. | 5780 (27.5) |  |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

14. Secondary Outcome: Phase 1a (Arm A and Arm B): Area Under the Plasma Concentration-Time From Time Zero Extrapolated to Infinity (AUC0-inf) of M3814 After Single Dose
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from the determination of the terminal first order (elimination) rate constant (lambda z). AUC0-inf = AUC0-t plus Clast pred/lambda z. Lambda z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 5 | 3 | 3 | 4 | 5 | 3 | 4 | 3 | 3
h*ng/mL
  Fraction Day 1: number analyzed (Participants) | 4 | 3 | 1 | 4 | 5 | 3 | 4 | 3 | 3
  Fraction Day 1 | 2480 (55.4) | 8780 (63.4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. | 16500 (61.8) | 1640 (82.9) | 4060 (77.3) | 17300 (108.6) | 1360 (48.8) | 3580 (59.6)
  Fraction Day 6: number analyzed (Participants) | 5 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 1200 (179.0) |  | 6890 (51.0) |  |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

15. Secondary Outcome: Phase 1a (Arm A and Arm B): Apparent Terminal Half Life (t1/2) of M3814 After Single Dose
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 was calculated by natural log 2 divided by Lambda z.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 5 | 3 | 3 | 4 | 5 | 3 | 4 | 3 | 3
hours
  Fraction Day 1: number analyzed (Participants) | 4 | 3 | 1 | 4 | 5 | 3 | 4 | 3 | 3
  Fraction Day 1 | 5.79 (47.6) | 7.81 (45.2) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. | 7.10 (27.9) | 3.20 (135.8) | 5.84 (34.6) | 5.83 (16.1) | 5.42 (79.8) | 5.85 (17.3)
  Fraction Day 6: number analyzed (Participants) | 5 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 6.57 (191.5) |  | 7.37 (79.1) |  |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

16. Secondary Outcome: Phase 1a (Arm A and Arm B): Total Body Clearance Following Oral Administration (CL/f) of M3814 After Single Dose
Description: The apparent total body clearance of study intervention following extravascular administration on FD1, taking into account the fraction of dose absorbed. CL/f = Dose oral (p.o.)/AUC0-inf. The predicted AUC0-inf should be used.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 5 | 3 | 4 | 3 | 3
liter per hour
  Fraction Day 1: number analyzed (Participants) | 4 | 3 | 1 | 3 | 5 | 3 | 4 | 3 | 3
  Fraction Day 1 | 40.4 (55.4) | 22.8 (63.4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. | 24.2 (61.8) | 60.9 (82.9) | 49.2 (77.3) | 17.3 (108.6) | 36.6 (48.9) | 27.9 (59.6)
  Fraction Day 6: number analyzed (Participants) | 5 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 83.2 (179.0) |  | 43.5 (51.0) |  |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

17. Secondary Outcome: Phase 1a (Arm A and Arm B): Apparent Volume of Distribution (Vz/f) of M3814 After Single Dose
Description: Apparent volume of distribution during the terminal phase following extravascular administration for M8891 was calculated. Vz/f = Dose/(AUC0-infinity multiply by Lambda z) following single dose. The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination. AUC(0- inf)=AUC0-t plus Clastpred/lambda z where Clastpred was last predicted concentration. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 1 and Fraction Day 6
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 5 | 3 | 4 | 3 | 3
liters
  Fraction Day 1: number analyzed (Participants) | 5 | 3 | 1 | 3 | 5 | 3 | 4 | 3 | 3
  Fraction Day 1 | 337 (64.5) | 257 (16.5) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. | 248 (45.6) | 280 (52.6) | 415 (61.2) | 146 (85.3) | 287 (48.0) | 235 (40.3)
  Fraction Day 6: number analyzed (Participants) | 5 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Fraction Day 6 | 790 (91.1) |  | 463 (41.4) |  |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  |  |

18. Secondary Outcome: Phase 1a (Arm A and Arm B): Maximum Plasma Concentration (Cmax) of M3814 After Multiple Dose
Description: Cmax was taken directly from the observed concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: Pharmacokinetic analysis set: all participants who received at least the first dose of the treatment (either M3814 or RT) and provided >= 3 valid post-dose concentration points within 6 hours (0-6 hours inclusive). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 2 | 0 | 4 | 5 | 2 | 4 | 7 | 3
ng/mL | 295 (97.1) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. |  | 1560 (84.8) | 575 (29.9) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 2020 (77.8) | 140 (60.3) | 392 (108.4)

19. Secondary Outcome: Phase 1a (Arm A and Arm B): Time to Reach Maximum Plasma Concentration (Tmax) of M3814 After Multiple Dose
Description: tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: as for outcome 18
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 2 | 0 | 4 | 5 | 2 | 4 | 7 | 3
hours | 2.00 [1.00 to 4.07] | NA [NA to NA] — Median and full range was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. |  | 2.18 [0.97 to 4.00] | 1.88 [0.50 to 2.08] | NA [NA to NA] — Median and full range was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 0.88 [0.75 to 1.00] | 2.00 [0.50 to 4.00] | 2.00 [0.63 to 2.00]

20. Secondary Outcome: Phase 1a (Arm A and Arm B): Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCtau) of M3814 After Multiple Dosing
Description: AUCtau was defined as area under the plasma concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: As per changes in planned analysis, the pharmacokinetic parameters (AUCtau) was not assessed.
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Phase 1a (Arm A and Arm B): Area Under the Plasma Concentration-Time From Time Zero Extrapolated to Infinity (AUC0-inf) of M3814 After Multiple Dose
Description: as for outcome 14
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: PK Analysis Set has been used here. The AUC-inf for peposertib cannot be calculated accurately when the sampling scheme is limited to 0-4 hours and the tmax ranges from 1 to 4 hours especially considering a half-life of 6 hours. Since the sampling scheme only covers 0-4 hours, the terminal elimination phase is not captured. As a result, it was not possible to calculate data for AUC0-inf because dosing interval was too small to have reliable results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 3 | 3 | 6 | 6 | 3 | 5 | 8 | 3
h*ng/mL | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description. | NA (NA) — Data could not be presented because of the reason mentioned in Analysis Population Description.

22. Secondary Outcome: Phase 1a (Arm A and Arm B): Apparent Terminal Half Life (t1/2) of M3814 After Multiple Dose
Description: as for outcome 15
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: Pharmacokinetic analysis set included all participants who received at least the first dose of the treatment (either M3814 or RT) and provided >= 3 valid post-dose concentration points within 6 hours (0-6 hours inclusive). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed"= participants evaluable for this outcome measure at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 3 | 1 | 0 | 1 | 2 | 0 | 4 | 2 | 1
hours | 8.37 (81.9) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation. | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. |  | 5.39 (27.3) | 3.30 (159.7) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

23. Secondary Outcome: Phase 1a (Arm A and Arm B): Oral Clearance in Plasma at Steady State (CLss/f) of M3814 After Multiple Dose
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: As per changes in planned analysis, the pharmacokinetic parameters (Clss/f) was not assessed.
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Phase 1a (Arm A and Arm B): Apparent Volume of Distribution at Steady-State (Vss/f) of M3814 After Multiple Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss/f after oral dose was influenced by the fraction absorbed.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 10
Population: As per changes in planned analysis, the pharmacokinetic parameters (Vss/f) was not assessed.
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Phase 1a (Arm A and Arm B): Accumulation Ratio of Area Under the Concentration-Time Curve (AUC) [Racc(AUC0-24)] of M3814 After Multiple Dose
Description: Accumulation ratio for AUC was calculated as AUC, after dosing on fraction Day 10 divided by AUC, after dosing on fraction Day 1 of cycle 1.
Time Frame: Pre-dose, 0.5, 1, 2, 4 and 24 hours post-dose on Fraction Day 1 and Fraction Day 10
Population: Pharmacokinetic analysis set included all participants who received at least the first dose of the treatment (either M3814 or RT) and provided >= 3 valid post-dose concentration points within 6 hours (0-6 hours inclusive). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 4 | 2 | 0 | 2 | 5 | 2 | 4 | 6 | 3
ratio | 1.38 (52.6) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. |  | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.44 (20.2) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 0.777 (55.0) | 0.922 (56.0) | 0.855 (60.7)

26. Secondary Outcome: Phase 1a (Arm A and Arm B): Accumulation Ratio of Cmax (Racc (Cmax) of M3814 After Multiple Dose
Description: Accumulation ratio for Cmax was calculated as Cmax, after dosing on fraction Day 10 divided by Cmax, after dosing on fraction Day 1 of cycle 1.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 1 and Fraction Day 10
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT
Number analyzed (Participants) | 7 | 2 | 0 | 4 | 5 | 2 | 3 | 7 | 3
ratio | 0.779 (108.1) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. |  | 0.871 (55.9) | 1.13 (50.9) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable participants were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 0.868 (58.9) | 0.816 (53.3) | 0.654 (61.7)

27. Secondary Outcome: Ancillary cPoP: Maximum Observed Plasma Concentration (Cmax) of M3814
Description: Cmax was taken directly from the observed concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 2
Population: Pharmacokinetic analysis set: all participants who received at least the first dose of the treatment (either M3814 or RT) and provided >= 3 valid post-dose concentration points within 6 hours (0-6 hours inclusive).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 3 | 3 | 1
ng/mL | 311 (148.2) | 504 (38.4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

28. Secondary Outcome: Ancillary cPoP: Time to Reach Maximum Plasma Concentration (Tmax) of M3814
Description: tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 2
Population: as for outcome 27
Measure: Median (Full Range); unit: hours
Groups:
- Ancillary cPOP: M3814 Capsule (400 mg) + RT: Participants with at least 2 (sub) cutaneous tumor/metastases of any type (at least 2 cm apart) with an indication for single high dose-palliative RT were included and received single oral dose of M3814 capsule at a dose of 400 mg on Day 2, prior 1.5 hours start of RT and a single high dose of RT (10-25 Gy) on Lesion 1 on Day 1 and on Lesion 2 on Day 2.
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 3 | 3 | 1
hours | 2.02 [2.02 to 2.42] | 1.03 [1.00 to 3.85] | NA [NA to NA] — Median and full range was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

29. Secondary Outcome: Ancillary cPoP: Area Under the Plasma Concentration-time Curve From Time Zero to 4 Hours (AUC0-4) of M3814
Description: AUC0-4hr is the area under the plasma concentration-time curve from time 0 to 4 hours post-dose. This is a measure of the average amount of study drug M3814 in the blood plasma over a period of 4 hours after the dose.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 2
Population: as for outcome 18
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 2 | 2 | 1
h*ng/mL | NA [NA to NA] — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

30. Secondary Outcome: Ancillary cPoP: Area Under the Plasma Concentration-time Curve From Time Zero to Last Sampling Time (Tlast) (AUC0-t) of M3814
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 2
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 3 | 3 | 1
h*ng/mL | 841 (172.4) | 1130 (47.2) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

31. Secondary Outcome: Ancillary cPoP: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/Dose) of M3814
Description: AUC0-t/Dose was defined as AUC from time of dosing to the time of the last measurable concentration divided by dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 2
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 3 | 3 | 1
h*ng/mL/mg | 8.41 (172.4) | 5.65 (47.2) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

32. Secondary Outcome: Ancillary cPoP: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to 4 Hours (AUC0-4)/Dose of M3814
Description: AUC0-4/Dose was defined as AUC from time of dosing to the time zero to 4 hours divided by dose.
Time Frame: Pre-dose, 0.5, 1, 2 and 4 hours post-dose on Fraction Day 2
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 2 | 2 | 1
h*ng/mL/mg | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

33. Secondary Outcome: Ancillary cPoP: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M3814
Description: Cmax/Dose was calculated as maximum observed plasma concentration obtained directly from the concentration versus time curve divided by dose. Cmax/dose was measured in nanogram per milliliter per milligram (ng/mL/mg).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6 hours post-dose on Fraction Day 2
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
Number analyzed (Participants) | 3 | 3 | 1
ng/mL/mg | 3.11 (148.2) | 2.52 (38.4) | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 1 collected value was not sufficient to calculate a reliable estimation.

ADVERSE EVENTS:
Time Frame: Time from first dose of study treatment up to long term safety follow-up period (Up to approximately 1 year)
Description: For Phase 1a (Arm A and Arm B): MedDRA Version 23.1 and for Ancillary clinical proof-of-principle (cPoP): MedDRA Version 22.1
Arm/Group | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT | Ancillary cPoP: M3814 Capsule (100 mg) + RT | Ancillary cPOP: M3814 Capsule (200 mg) + RT | Ancillary cPOP: M3814 Capsule (400 mg) + RT
All-Cause Mortality (participants affected / at risk) | 4/7 | 2/3 | 2/3 | 6/6 | 3/6 | 2/3 | 3/6 | 1/8 | 1/3 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/3 | 2/3 | 2/6 | 1/6 | 0/3 | 3/6 | 2/8 | 1/3 | 1/3 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 2/3 | 6/6 | 6/6 | 3/3 | 6/6 | 8/8 | 3/3 | 2/3 | 3/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT (N=7) | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT (N=3) | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT (N=3) | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT (N=6) | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT (N=6) | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT (N=3) | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT (N=6) | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT (N=8) | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT (N=3) | Ancillary cPoP: M3814 Capsule (100 mg) + RT (N=3) | Ancillary cPOP: M3814 Capsule (200 mg) + RT (N=3) | Ancillary cPOP: M3814 Capsule (400 mg) + RT (N=1)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a (Arm A): M3814 Capsule (100 mg) + RT (N=7) | Phase 1a (Arm A): M3814 Capsule (200 mg) + RT (N=3) | Phase 1a (Arm A): M3814 Capsule (300 mg) + RT (N=3) | Phase 1a (Arm A): M3814 Capsule (400 mg) + RT (N=6) | Phase 1a (Arm A): M3814 Tablet (100 mg) + RT (N=6) | Phase 1a (Arm A): M3814 Tablet (200 mg) + RT (N=3) | Phase 1a (Arm A): M3814 Tablet (300 mg) + RT (N=6) | Phase 1a (Arm B): M3814 Capsule (50 mg) + CRT (N=8) | Phase 1a (Arm B): M3814 Tablet (100 mg) + CRT (N=3) | Ancillary cPoP: M3814 Capsule (100 mg) + RT (N=3) | Ancillary cPOP: M3814 Capsule (200 mg) + RT (N=3) | Ancillary cPOP: M3814 Capsule (400 mg) + RT (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 4 | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 5 | 2 | 1 | 2 | 6 | 2 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 2 | 0 | 4 | 7 | 3 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue movement disturbance (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 3 | 3 | 2 | 0 | 0 | 0
Application site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 2 | 0 | 5 | 2 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation dysphagia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 4 | 5 | 1 | 4 | 6 | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 5 | 2 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular pain (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT02516813/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT02516813/SAP_001.pdf